CLINICAL TRIAL: NCT04900688
Title: First Clinical Evaluation of the New Flexible Disposable Ureteroscope (LithoVue Elite): A Multicenter Single-arm Prospective Trial
Brief Title: Prospective Evaluation of the LithoVue Elite Ureteroscope
Acronym: LVE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Collaborators: University of British Columbia (Other); Western University, Canada (Other); Université de Montréal (Other); University of Saskatchewan (Other); Laval University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MP-02-2022-9937
Record Dates: First submitted 2021-05-20; First posted 2021-05-25 (Actual); Last update posted 2024-06-07 (Actual); Status verified 2024-06

CONDITIONS: Kidney Stone
Keywords: renal stone, ureteroscopy, laser lithotrypsy, ureteroscope
MeSH Terms: conditions — Kidney Calculi; Nephrolithiasis

STUDY DESIGN:
Intervention Model Description: Single arm multicenter study looking at real world results of ureteroscopy with the new digital flexible ureteroscope.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ureteroscopy (URS) with the LithoVue Elite disposable flexible ureteroscope (Other): Ureteroscopy will be done using the LithoVue Elite disposable flexible ureteroscope instead of the satandard ureteroscope
  Interventions: Device: LithoVue Elite

INTERVENTIONS:
Device: LithoVue Elite — LithoVue Elite is a disposable flexible ureteroscope that offer novel pressure sensory capacity

SUMMARY:
Flexible ureteroscopy has become the main surgical treatment for kidney stone disease. The procedure uses many types of ureteroscopes (disposable and non-disposable). Currently we are using the LithoVue Single-Use Digital Flexible Ureteroscope. The Health Canada approved LithoVue Elite disposable flexible ureteroscope will now offer novel pressure sensory capacity. In order to evaluate the new ureteroscopy we will be conducting a prospective multi-institution study in order to determine the main features, capacity and abilities of the new scope. We will evaluate the impact of intra renal pressure on pain, quality of life and possible infectious complications.

DETAILED DESCRIPTION:
This is a single arm multicenter study looking at real world results of ureteroscopy with the new digital flexible ureteroscope LVE. The study will involve 6 participating institutions. Each site will be in charge of recruiting 25 participants for a total of 150 participants.

Hypothesis:

1. The single-use flexible ureteroscope (Lithovue Elite) will provide equivalent overall performance to a standard-of-care reusable or disposable ureteroscope as determined by:

   * Stone-free rate following ureteroscopy at 4-8 weeks post-procedure
   * Equivalent adjunctive procedures in the postoperative period
   * Intraoperative assessment parameters will show no difference between the Lithovue Elite scope and other standard-of-care ureteroscopes
2. Elevated intrarenal pressures during ureteroscopes will result in:

   * Higher post-operative pain intensity as documented in the Brief Pain Inventory-BPI
   * Lower quality of life as reflected via Wisconsin Stone Quality of Life Questionnaire scores
   * Higher rates of infections complications
   * Changes in neutrophil gelatinase-associated lipocalin (NGAL) from baseline

Procedures:

Patients who will undergo ureteroscopy and laser lithotripsy will be screened for eligibility. The stone burden needs to be less than 20 mm in total to be eligible. Patients with a nephrostomy tube are ineligible as the nephrostomy tube may affect the intraoperative renal pressure. Patients undergoing bilateral ureteroscopy are eligible to participate.

Eligible patients will be approached to participate in the study, their consent will be obtained and each participant will be assigned an identification number to code his/her data. Patients will undergo standard-of-care ureteroscopy under anesthesia specific to the investigator's site.

Preoperatively, patients who have an indication to undergo ureteroscopy will have imaging and fill out a WISQOL and BPI questionnaire at baseline. Baseline urine analysis is required and culture if indicated as per standard of care. Bloodwork is performed as per institutional standard of care. In addition, a urine sample will be obtained and stored (-20C) for NGAL measurement. The standard-of-care at each site will be used for antibiotics and whether the procedure is performed as an outpatient procedure or if the patient is admitted to the hospital post-operatively The day of surgery, the ureteroscopy will be performed using the new digital flexible ureteroscope LithoVue Elite (LVE). It will be carried out as per the surgeon's preference as to the use of a safety guidewire, use of ureteral access sheath (UAS), basketing stones or dusting, type of laser used, and laser settings. The irrigation used will be recorded and used as per the surgeon's preference. The pressure readings from LVE will be recorded. A decision on whether to leave a stent and its indwelling time is left up to the surgeon. Stone (s) will be sent for laboratory analysis.

In the recovery room after the procedure, the patient will have their Quick Sequential Organ Failure Assessment Score (QSOFA) score measured (systolic blood pressure, mentation status (GCS), and respiratory rate) as well as complete the BPI. In addition, a urine sample will be obtained and stored (-20C) for NGAL measurement as well as any other laboratory tests requested by the investigator. Postoperative antibiotics, analgesics (e.g. Tylenol, NSAID, +/- opioid) and discharge medication (e.g. NSAIDS, Opioids, Anticholinergics, Alpha blockers) prescriptions are left to the discretion of surgeon and will be recorded.

Within 1-2 weeks, participants who have a stent will come to the hospital for stent removal. Stents can be removed in any fashion (tether string or cystoscopy), this decision is left up to the surgeon. Participants who have no stent in place might have an in-person or remote follow-up depending on COVID 19 restrictions. Participants will have to also complete the BPI and WISQOL.

Within 4-8 weeks postoperatively, patients will undergo standard of care imaging with either a combination of KUB x-ray and renal-bladder ultrasound or a low-dose CT scan. The choice of modality will be left to the surgeon discretion depending on institutional standards, surgeon preference and stone type. The stone free rate will be recorded based on imaging results. Participants will complete the BPI and WISQOL. The patient will have completed the study.

Study visits and measurements:

Preoperative visit (V0) : During this visit we will record:

1. Demographics data: sex, date of birth (month and year), date of surgery, age, height, weight, BMI, comorbidities, Charlson Comorbidity Index.
2. Preoperative data: Stent preop, blood work, urine analysis, urine culture, treatment of UTI, baseline NGAL measurement, imaging modality, medication.
3. Stone- related data based on imaging results: Number of stones, Stone location, size (length, width, height), volume, DICOM Volume and density (HU)
4. Patient reported outcomes: participants will complete the WisQOL, and BPI (baseline).

Day of surgery visit (V1) : During this visit we will perform ureteroscopy with laser lithotripsy per usual and collect the following data:

1. Intraoperative data: ASA score, date and duration of surgery, type of anesthesia, type of procedure, use of Ureteral Access Sheath (UAS), Safety Guide Wire (SGW), Laser and their related information (type, size, settings), surgical technique (basketing or dusting), irrigation related information, intraoperative pressure measurement, use of stent and strings, perioperative antibiotics, intraoperative complications, ability to navigate all areas of the kidney and complete the entire case using one-single use ureteroscope.
2. Recovery room data: QSOFA, NGAL measurement, postoperative analgesics, discharge medication and postoperative antibiotics.
3. Patient reported outcomes: At discharge from the recovery room participants will complete the BPI.

Postoperative visit (V2): Within 1-2 weeks we will remove the stent and record;

1. Postoperative data: Date of stent removal and stent indwelling time when applicable
2. Patient reported outcomes: Participants will complete the WisQOL and BPI

Postoperative visit (V3): Within 4-8 weeks postoperatively, patients will undergo standard of care imaging. During this visit we will record:

1. Postoperative information: Postoperative imaging modality and Stone-free Rate (SFR), type of stone (s) based on stone's laboratory analysis and 30 days-postoperative complications.
2. Patient reported outcomes: Participants will complete the WisQOL and BPI.

Additional variables collected allowing ancillary studies. Medical charts of participants and surgical protocol will be reviewed to collect the information needed for this study.

Data collection, management, storage and conservation:

Data collection and management:

A urine sample will be drawn for NGAL measurement at V0 and V1. The sample will be stored in a freezer at -20C at each participating center. Analysis of urine samples will done at the University of British Columbia's laboratory in Vancouver, shipment of samples for analysis will be done once, at the end of the study. Samples will be destroyed after analysis.

Redcap database will be used for data collection. Each participating center will be provided an access to CHUM's REDCap to enter all data requested during the study (demographic data as well as patient reported outcomes, clinical data, imaging and laboratory results). Patient reported outcomes-related questionnaires can be sent via REDCap powered emails to be completed online or given to participants in paper form depending on the site's preference.

Data storage and conservation:

Nominal data as well as the file that links identification information with the code assigned to each participant will be stored and kept at each participating institution as required by each institution's Research Ethics Board.

No identification data will be stored on REDCap, except the e-mail address of participants for the sites that will use REDCap powered emails to send the questionnaires to participants. Data collected and stored on REDCap will be coded and the e-mail address of participants will be removed at the time of data extraction for analysis.

Only the members of the Central Coordinating Research Team at the CHUM who are involved in the study, the local coordinators at participating sites and the REDCap data manager at the CHUM will have access to data stored on REDCap. The data collected using REDCap will be hosted on secure CHUM servers.

There is no blinding during this study and it is not an interventional trial so emergency access to the database is not necessary for patient care. It is an observational trial and measuring patient reported outcomes. At the end of the study, data collected via REDCap will be downloaded for analysis, stored on the network drive of Dr. Naeem Bhojani at the CHUM and kept for 10 years.

Ethical considerations:

The procedures of this study fall within standard-of-care, and as such all prospective patients to be enrolled in this study will receive the same care whether they are included in the study or not. These patients may withdraw from the study at any time without any negative consequences to the medical care, education, or other services to which they are entitled or are presently receiving.

Intrarenal pressure measurements during the study ureteroscopy procedure is not part of the standard of care and is done for research purposes only. There is no additional risk to the patient when monitoring this pressure and patients will be informed of this during the informed consent process.

NGAL measurement is a measurement that is not part of standard of care, at the preoperative visit urine analysis are done as part of usual care, the medical staff will ask patients for an additional urine sample to be stored (-20C) for NGAL measurement. Right after their ureteroscopy (V1) while in the recovery room, no urine sample is drawn as part of standard care, we will ask participants to provide a urine sample exclusively for NGAL measurement but participants will be informed of this. No more NGAL measurements are required as part of study procedures.

Approached participants will be asked to provide their consent. Paper or electronic consent might be used depending on participating site preferences and Research Ethics Board requirements. Electronic consent might be obtained via REDCap or other means/platforms as authorized by each participating site Research Ethics Boards.

Data collected during this study will be kept for 10 years. The results will be presented at conferences and published in journals; however, precautions will be taken to ensure that at the time of dissemination, the study participants will not be identifiable.

Funding:

This is an investigator-initiated trial and there is no funding for this study.

Conflict of interest:

Although this is an investigator-initiated study, it should be noted that the principal investigator (Dr Naeem Bhojani) and the Co-Principal investigator (Dr. Ben Chew) are consultants for Boston Scientific, the manufacturer of the LithoVue Elite disposable flexible ureteroscope under evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Patient scheduled for ureteroscopy and laser lithotripsy
* Non-obstructing renal stone 2 cm total stone diameter (if multiple stones, then sum of maximum diameters) or less undergoing flexible ureteroscopy
* age > 18 years

Exclusion Criteria:

* age < 18 years
* pregnancy status =positive
* indwelling nephrostomy tube
* severe hydronephrosis that in the opinion of the investigator, will make it challenging to make the patient stone free
* renal anomalies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2023-01-16 (Actual); Primary Completion 2025-03-15 (Estimated); Study Completion 2025-09-15 (Estimated)

PRIMARY OUTCOMES:
WISQOL | At baseline, 1-2 weeks after surgery and 4-8 weeks after surgery
  Change in quality of Life of patients living with kidney stones as assessed by the Winsconsin Stone Quality Of Life questionnaire

SECONDARY OUTCOMES:
BPI | at baseline, in the recovery room after surgery, 1-2 weeks after surgery and 4-8 weeks after surgery
  Change in pain intensity as assessed by the Brief Pain Inventory Questionnaire (BPI)
Stone free rate | 4-8 weeks after surgery
  Stone free rate as assessed by imaging
Infectious Complications | at 30 days after surgery
  Postoperative infectious Complications as assessed by the healthcare provider
Complications | at 30 days after surgery
  Postoperative complications as assessed by the healthcare provider
Change in neutrophil gelatinase-associated lipocalin (NGAL) from baseline | at baseline and in the recovery room after surgery
  NGAL is a marker of kidney injury. NGAL measurement will de done on a urine sample

CONTACTS AND LOCATIONS:
Overall Officials: Naeem Dr Bhojani, MD, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (6):
- Canada (6):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Western University, London, Ontario
  - Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec
  - Hôpital Maisonneuve-Rosemont (HMR), Montreal East, Quebec
  - CHU de Québec-Université Laval, Québec, Quebec
  - University of Saskatchewan, Saskatoon, Saskatchewan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Benli E, Ayyildiz SN, Cirrik S, Noyan T, Ayyildiz A, Cirakoglu A. Early term effect of ureterorenoscopy (URS) on the Kidney: research measuring NGAL, KIM-1, FABP and CYS C levels in urine. Int Braz J Urol. 2017 Sep-Oct;43(5):887-895. doi: 10.1590/S1677-5538.IBJU.2016.0638. PMID 28792192
- [Background] Fahmy N, Sener A, Sabbisetti V, Nott L, Lang RM, Welk BK, Mendez-Probst CE, MacPhee RA, VanEerdewijk S, Cadieux PA, Bonventre JV, Razvi H. Urinary expression of novel tissue markers of kidney injury after ureteroscopy, shockwave lithotripsy, and in normal healthy controls. J Endourol. 2013 Dec;27(12):1455-62. doi: 10.1089/end.2013.0188. Epub 2013 Nov 1. PMID 24180435
- [Background] Penniston KL, Antonelli JA, Viprakasit DP, Averch TD, Sivalingam S, Sur RL, Pais VM Jr, Chew BH, Bird VG, Nakada SY. Validation and Reliability of the Wisconsin Stone Quality of Life Questionnaire. J Urol. 2017 May;197(5):1280-1288. doi: 10.1016/j.juro.2016.11.097. Epub 2016 Nov 23. PMID 27889419